CLINICAL TRIAL: NCT06345027
Title: Chimeric Antigen Receptor Treatment Targeting CD70 (SEVENTY)
Acronym: CASEY
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Bilal Omer, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-53163 CASEY
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, B-cell; Leukemia, T-Cell
Keywords: Leukemia; Acute myeloid; B cell; T cell; Blood cancer; Lymph gland cancer; CD70.CAR T-cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, B-Cell; Leukemia, T-Cell; Leukemia; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm A (Experimental): Patients will initially be consented for procurement of blood for generation of the transduced T-cells.
  Three dose levels will be evaluated and a possible dose level -1 in case of unexpected toxicity at dose level 1. Each patient will receive one T cell infusion.
  Interventions: Biological: Treatment Arm A

INTERVENTIONS:
Biological: Treatment Arm A — Each patient will receive one T cell infusion.
  CD70.CAR Dose Levels / Cell Dose (transduced cells):
  Dose Level -1: 3 x 10^5 cells/kg Dose Level 1 (starting dose level): 1 x 10^6 cells/kg Dose Level 2: 3 x 10^6 cells/kg Dose Level 3: 1 x 10^7 cells/kg
  *First three patients treated on the study will be adults 18 years of age or older.

SUMMARY:
This study is for patients who have a type of blood cancer that expresses the protein CD70, which includes acute myeloid leukemia (AML), T-cell leukemia or B-cell leukemia (and the leukemia has come back or has not gone away after standard of care treatment).

As there are limited or no remaining standard treatments available to treat this cancer, subjects are being asked to volunteer to be in a gene transfer research study using special immune cells to create a specialized immune cell that will recognize a protein called CD70 that is expressed on the outside surface of the leukemia cells in a subject's body.

The body has different ways of fighting infection and disease. No one way seems perfect for fighting cancers. This research study combines different ways of fighting disease by using T cells and "arming" them to recognize a specific protein on cancer cells. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells including tumor cells. T cells by themselves have been used to treat patients with cancers and have shown promise, but have not been strong enough to cure most patients.

T lymphocytes can kill tumor cells but there normally are not enough of them to kill all the tumor cells. Some researchers have taken T cells from a person's blood, grown more of them in the laboratory and then given them back to the person.

The protein used in this study is called anti-CD70. It has been developed from human CD27 on normal T cells, since it is the natural binding partner that can connect with CD70. This anti-CD70 protein sticks to leukemia cells when it binds to CD70. CD70 binders have been used to treat people with leukemia. For this study, anti-CD70 has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor or "CAR T cell". The doctors then made another change to cause these T cells to kill any cell that has CD70. This causes the "CAR T cells" to kill blood cancer cells which are confirmed to have CD70.

In the laboratory, investigators have found that T cells work better if there are proteins added which stimulate T cells. The anti-CD70 (CD27) protein is unique because it can bind to CD70 on leukemia cells but also stimulates the T cells that express it. Adding the CD27 makes the cells grow better and may help them to last longer in the body, thus giving the cells a better chance of killing the leukemia cells.

These CD70 "CAR" T cells are investigational products not approved by the Food and Drug Administration.

The purpose of this study is to find a dose of CAR T cells that is safe, to learn what the side effects are and to see whether this therapy might help people with leukemia.

DETAILED DESCRIPTION:
Patients will be enrolled to this study in two treatment groups: C7R-EBVSTs without lymphodepletion (Group A) and C7R-EBVSTs with lymphodepletion (Group B). The investigators will enroll patients into group B if limited expansion and clinical effectiveness is seen in Group A.

Patients will give blood to make C7R EBV T cells. These cells will be kept frozen until they are given to the patient.

The lines are made using a special process. To make the VSTs donor cells are mixed with small pieces of proteins, called peptides that are identical to proteins from EBV. First unwanted cells are separated from the donor blood. The unwanted cells have CD45RA on their surface and can be identified and removed from the product leaving behind only the T cells that contain a small number of VSTs. The cells are then stimulated with the peptides to make them grow. After about 9 days the growth of the VSTs starts to slow down and they are stimulated a second time (and possibly a third) with peptides together with cells from the donor that have been modified to help train the T cells to kill cells that are infected with EBV as well as a cell line (called ULCL) that helps the T-cells to grow. ULCL is made by infecting lymphocytes with EBV that has been made non-infectious by deleting a part of its DNA. ULCL is irradiated before use so that it cannot grow. Once enough VSTs are made they are frozen and tested to make sure they can recognize virus infected cells but not normal cells.

To get the C7R to be made by the T-cell, a gene is inserted into the T-cell. This is done using certain parts of a virus (known as a retrovirus). A retrovirus is a type of virus that inserts a copy of its own genetic material into the DNA of a different host cell. The retrovirus can carry the gene into the T cells. Patients that have received cells with a new gene in them will be followed for a total of 15 years in order to see if there are any long term side effects of gene transfer. Gene transfer is the insertion of genetic material into a cell.

Patients that enroll on this study will be assigned a dose of C7 R EBV T cells. The assigned dose of cells is based on body weight and height. In Group A, in this study patients will receive the C7 R EBV T cells. If in Group B, along with the C7R EBV T cells, patients will and may also receive cyclophosphamide and fludarabine. These two drugs are standard chemotherapy medicines and may be given before the T cells to make space in the blood for the T cells to grow after the patient has received them.

If in Group B, patients may receive cyclophosphamide and fludarabine, these drugs will be given intravenously (through an i.v. needle inserted in the vein or the central line) for 2 days and then fludarabine alone on the third day (Day -4, -3, -2) before the infusion. On Day 0, patients will be given an injection of C7 R EBV T cells into the vein through an IV line at the assigned dose.

Before receiving the T cell infusion, patients may be given a dose of Benadryl (diphenhydramine) and Tylenol (acetaminophen). The infusion will take between 1 and 10 minutes. Patients will be monitored in the clinic or hospital for about 2 hours. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital. Patients should plan to stay in Houston for at least 2 weeks after the infusion to be monitored for side effects.

Patients will have follow-up visits with the clinic after the infusion (at scheduled visits weeks 2 and 6, and nursing follow up at weeks 1, 2, 4 and 6 after the infusion, and at months 3, 6, 9, and 12 after the infusion. The patients will also have nursing follow up annually for the next 15 years, and scheduled disease evaluations after the T-cell injection (at week 6 +/- 2 weeks after the infusion and then as clinically needed).

After disease re-evaluation, if the disease has not gotten worse, or if in the future it seems that patients might benefit and have not had a severe side effect caused by the infusion of the C7R EBV T cells, the patients may be eligible to receive one additional dose of the T cells. The dose will be at the same dose level as the first infusion and separated by at least 4 weeks to make sure there are no severe side effects between infusions. Patients that receive an additional dose of C7R EBV T-cells, should plan to stay in Houston for at least 2 weeks after the infusion to be monitored for side effects.

Medical tests before treatment--

Before being treated, patients receive a series of standard medical tests:

1. Physical exam
2. Blood tests to measure blood cells, kidney and liver function
3. Measurements of the tumor by routine imaging studies. Imaging studies that have been used in the past will be used to best assess the tumor (Computer Tomogram (CT) or Magnetic Resonance Imaging (MRI), and Positron Emission Tomography (PET/CT) and/or Bone Scan).

Medical tests during and after treatment--

Patients will receive standard medical tests while receiving the infusions and afterwards:

1. Physical exams
2. Blood tests to measure blood cells, kidney and liver function
3. Measurements of the tumor by routine imaging studies approximately 6 weeks after the infusion.
4. Tumor biopsy of an accessible tumor between 2-4 weeks after the infusion and as clinically indicated thereafter.

To learn more about the way the C7R EBV T cells are working and how long they last in the body, an extra amount of blood will be obtained on the day that chemotherapy starts, on the day of the T-cell infusion(s) and at the end of the T-cell infusion(s). Blood will also be obtained at 1, 2, 4, 6 weeks after the T-cell infusion(s) and every 3 months for the 1st year. Blood will then be obtained annually for the next 15 years and possibly at additional time points. The amount of blood taken will be based on weight with up to a maximum of 60 mL (12 teaspoons) of blood to be obtained at any one time. For children, the total amount of blood drawn will not be more than 3 mL (less than 1 teaspoon) per 2 lbs (1 kg) of body weight on any one day. This volume is considered safe, but may be decreased if the patient is anemic (have a low red blood cell count).

ELIGIBILITY:
Procurement Inclusion Criteria:

1. Diagnosis of primary refractory or relapsed Acute Myeloid Leukemia (AML) with the exception of acute promyelocytic leukemia (APL). Patients with targetable mutations should have failed or be ineligible for targeted therapies (e.g. FLT3 inhibitors, IDH inhibitors or anti-CD33 drug conjugate)

   OR

   Patients with other relapsed or refractory CD70+ leukemia that would be considered an indication for allogeneic Hematopoietic Stem Cell Transplant (HSCT) if remission can be achieved. (CD19+ leukemia only: Patients must have failed or be ineligible to receive commercial CD19.CAR T cell treatments.)

   Primary refractory or resistant disease, for purposes of procurement, defined as not achieving complete remission (CR) (i.e., a remaining blast count of 5% or more) after 1 to 2 cycles of intense induction therapy.

   Relapse is defined as (1) hematologic relapse after complete remission based on bone marrow blasts >=5%, or reappearance of blasts in the blood, or development of extramedullary disease; (2) molecular relapse after minimal residual disease (MRD) negative, complete remission based on reoccurrence of MRD as assessed by RT-qPCR or by multi-parametric flow cytometry (MFC)
2. CD70 positive leukemia with at least 26% CD70+ blasts by flow cytometry or immunohistochemistry (staining can be pending at time of procurement)
3. Age ≤75 years. NOTE: The first three (3) patients treated on the study will be adults (≥18 years of age)
4. Hemoglobin ≥ 7.0 g/dL (can be transfused)
5. If apheresis required to collect blood

   * PT and aPTT <1.5x ULN
   * Serum Creatinine < 2 x ULN
   * AST < 5 x ULN
6. Informed consent

Procurement Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL)
2. Active infection (bacterial, fungal, or viral) requiring ongoing treatment without improvement.
3. Known active infection with HIV or HTLV (collected blood will be sent for HIV/HTLV testing, separate testing prior to procurement not required). Patients with HIV are eligible if viral load is undetectable on therapy and CD4 count is >350 mm3.
4. Active second cancer (except non-melanoma skin cancer or in situ breast cancer or cervical cancer) or other cancer treated ≤ 2 years prior to enrollment
5. Ongoing treatment with immune suppression for prophylaxis/treatment of GVHD including high dose steroids (e.g. prednisone equivalent > 0.5 mg/kg/day)

Treatment Inclusion Criteria:

1. Diagnosis of primary refractory or relapsed Acute Myeloid Leukemia (AML) with the exception of acute promyelocytic leukemia (APL) Patients with targetable mutations should have failed or be ineligible for targeted therapies (e.g. FLT3 inhibitors, IDH inhibitors, or anti-CD33 drug conjugate).

   OR

   Patients with other relapsed or refractory CD70+ hematological leukemias that would be considered an indication for allogeneic Hematopoietic Stem Cell Transplant (HSCT) if remission can be achieved. Patients with CD19+ malignancies must have failed or be ineligible to receive commercial CD19.CAR T cell treatments.

   Primary refractory or resistant disease as defined by not achieving complete remission (CR) (i.e., a remaining blast count of 5% or more) after 1 to 2 cycles of intense induction therapy. Patients with no reduction in blast count after the first cycle or with p53 mutations without CR after the first cycle of intense induction therapy are also considered primary refractory.

   Relapse is defined as (1) hematologic relapse after complete remission based on bone marrow blasts >=5%, or reappearance of blasts in the blood, or development of extramedullary disease; (2) molecular relapse after minimal residual disease (MRD) negative, complete remission based on reoccurrence of MRD as assessed by RT-qPCR or by multi-parametric flow cytometry (MFC)
2. Confirmation from the patient's primary physician team of a suitable allogeneic hematopoietic stem cell transplant (HSCT) donor. OR Documentation that patient declines a potential subsequent HSCT)
3. CD70 positive leukemia with at least 26% CD70+ cells by flow cytometry or immunohistochemistry (tissue)
4. No systemic chemotherapy at least 2 weeks prior to treatment on study and must be recovered from all acute toxic effects of prior chemotherapy at time of treatment.
5. Age ≤ 75 years. NOTE: The first three (3) patients treated on the study should be adults (≥18 years of age). Thereafter, a thorough review of the safety data will be performed and submitted to the FDA for approval prior to enrolling pediatric patients.
6. Hemoglobin ≥ 7.0 g/dL (can be transfused)
7. Total bilirubin < 3 times the upper limit of normal
8. AST/ALT < 5 times the upper limit of normal
9. Estimated GFR ≥ 60ml/min
10. Pulse oximetry of > 90% on room air
11. Karnofsky/Lansky score of ≥ 60%
12. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. Male partner should use a condom
13. Informed consent obtained

Treatment Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL)
2. Currently receiving any investigational agents or received any tumor vaccines within the previous 6 weeks.
3. Pregnant or lactating.
4. Uncontrolled infection with HIV, or HTLV. Patients with HIV are eligible if viral load is undetectable on therapy and CD4 count is >350 mm3.
5. Clinically significant bacterial, fungal, or viral infection requiring ongoing therapy without improvement.
6. Cardiac abnormalities: Cardiac echocardiography with LVEF<50%; Cardiac dysfunction NYHA III or IV; Clinically significant pericardial effusion. Confirmation of absence of these conditions within 6 months of treatment.
7. Presence of CNS disease: Defined as detectable cerebrospinal blast cells in a sample of CSF with ≥ 5 WBCs per mm3 or known CNS tumors/chloromas (repeat spinal tap within 4 weeks only required for leukemia patients with known CNS disease)
8. Use of serotherapy with Campath or Anti-Thymocyte Globulin (ATG) within the last 28 days
9. Use of Donor Lymphocyte Infusion (DLI) or other cellular therapy product within 28 days
10. Acute GVHD ≥ Grade 2 or moderate to severe (formerly extensive) chronic GVHD
11. High dose steroids >1 mg/kg within preceding 5 days or currently receiving >0.5mg/kg/day prednisone equivalent
12. Hyperleukocytosis (WBC ≥ 50K) or rapidly progressive disease that in the estimation of the investigator would compromise the ability of the patient to complete the initial 6 weeks of the study

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2042-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) rate | Time Frame 4 weeks post infusion
  1. Dose-limiting toxicity (CTCAE v5.0) is defined as any grade 3 or 4 non-hematologic toxicities (including allergic reactions and ICANS) that fails to return to Grade 2 within 72 hours or any grade 5 toxicity (additional assessment criteria may apply).

SECONDARY OUTCOMES:
Overall Response Rate | Time Frame 4 weeks post infusion
  1. Response rate by International Working Group Criteria for AML and disease specific response criteria for patients with other hematological malignancies.
  The response rate for AML is calculated as the overall complete response rate (CRMRD- + CR + CRi)

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Omer, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas